CLINICAL TRIAL: NCT01361490
Title: Rehabilitating Overweight People Back to Working Life
Acronym: ARRO
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: RSSO 2010/3
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obesity may have implications on the individual's participation in working life through different mechanisms such as comorbidity and loss of functional level. The investigators also know that when exiting the working force, it is difficult to get back later. As rehabilitation back to working life is often not a very focused aim with weight loss treatment, this study sets this as a primary aim by involvement in a 4 week stay at a rehabilitation clinic followed by 48 weeks work practice programme at one of three different companies.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-47
* 19-67 years

Exclusion Criteria:

* Pregnancy
* Significant reduced physical function
* Drug use
* Serious mental illness

Ages: 19 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese people where the obesity is the reason they are not actively taking part in working life.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Participation in working life | 4 years

SECONDARY OUTCOMES:
Body weight | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Muritunet Rehabiliteringssenter, Valldal, Norway